CLINICAL TRIAL: NCT05477823
Title: Pilot Study to Identify Radiogenomic Biomarkers to Predict Early Treatment Response to Androgen Deprivation Therapy and Radiation Therapy in High Risk Prostate Cancer
Brief Title: Imaging and Genomic Biomarkers to Predict Response in Prostate Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2022-0493; 2022-0493 (Other: UW Madison); Protocol version 9/5/2025 (Other: UW Madison); A533300 (Other: UW Madison); SMPH/HUMAN ONCOLOGY/HUMAN ONCO (Other: UW Madison); UW20099 (Other: OnCore ID)
Record Dates: First submitted 2022-07-21; First posted 2022-07-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- EBRT + BTX + ADT, PET and MRI (Experimental): Standard of care EBRT + BTX + ADT, with mid-treatment PET and MRI (or PET and CT) scans for research.
  Interventions: Radiation: External beam radiation therapy; Radiation: Prostate brachytherapy boost; Drug: Androgen deprivation therapy; Diagnostic Test: Positron emission tomography (PET)/magnetic resonance imaging (MRI)

INTERVENTIONS:
Radiation: External beam radiation therapy — Standard of care EBRT
Radiation: Prostate brachytherapy boost — Standard of care BTX
Drug: Androgen deprivation therapy — Standard of care ADT
Diagnostic Test: Positron emission tomography (PET)/magnetic resonance imaging (MRI) — Pelvic PET scanning with tracer will take approximately 45 minutes. This will be followed by the injection of a contrast agent followed by whole body PET/MRI scanning which will take approximately 30 minutes.

SUMMARY:
The purpose of this study is to evaluate the imaging and gene expression biomarkers in prostate cancer. Participants have high-risk prostate cancer and have indicated they will undergo external beam radiation therapy, brachytherapy, and androgen deprivation therapy (EBRT+BTX+ADT). Participants can expect to be in this study for up to 5 years.

DETAILED DESCRIPTION:
This is a pilot study to prospectively investigate potential predictive imaging and genomic biomarkers for patients with high-risk prostate cancer treated with standard of care EBRT + BTX + ADT. The primary imaging modalities that will be evaluated will be PSMA positron emission tomography (PET) and multi-parametric magnetic resonance imaging (MRI). Pre-treatment PET/MRI scans will also be obtained as part of standard of care prior to study enrollment. Response will be assessed on a mid-treatment PET/MRI scan obtained for research purposes after completion of EBRT but prior to brachytherapy boost. PET/CT (computerized tomography) may be used instead if PET/MRI is not technically possible. Imaging response will be compared to pathology from image-directed prostate biopsies taken at the time of the brachytherapy boost. The primary genomic marker that will be evaluated is a clinically available gene-expression array, Decipher, that will be obtained as part of standard of care prior to study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Histologically confirmed adenocarcinoma of the prostate
* Cancer classified as high-risk or very high-risk by National Comprehensive Cancer Network (NCCN) criteria: Grade group ≥4, PSA >20, or primary tumor stage ≥T3a
* ECOG performance status 0-1
* Agreed to undergo EBRT, high dose rate (HDR) brachytherapy boost, and 6-36 months of ADT as part of standard of care therapy prior to study enrollment
* Able to undergo a HDR brachytherapy implant: Pre-radiation IPSS score ≤20 with or without medical management; prostate ≤60 cc as measured by MRI or ultrasound; no prior trans-urethral resection of prostate (TURP); and, median lobe extending into the bladder <1 cm
* No prior or concurrent malignancy unless disease-free for at least 5 years

Exclusion Criteria:

* Evidence of regional or distant metastatic disease on pre-treatment bone scan, pelvic MRI, and/or CT of the abdomen/pelvis
* Prior pelvic radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Imaging markers for mid-treatment response | Mid-treatment (approximately 3 months into treatment)
  Evaluate prostate specific membrane antigen (PSMA) PET/MRI for imaging biomarkers that predict mid-treatment response to ADT and EBRT to identify participants at risk for poor response to radiation therapy and ADT.

SECONDARY OUTCOMES:
Genomic signatures correlated with imaging response | Baseline and mid-treatment (approximately 3 months into treatment)
  Determine if the Decipher and PORTOS genomic scores (high vs low) and basal/luminal genomic subtypes are correlated with change in PSMA standardized uptake value (SUV) pre-to-mid-treatment.
Establish a correlation between PET imaging response and pathologic response | Baseline and mid-treatment (approximately 3 months into treatment)
  PET images will be assessed for response using change in SUV in order to establish a correlation between imaging response and pathologic response to ADT and EBRT on a lesion-by-lesion basis. Pathologic response will be evaluated considering change in percent core involvement, prostate cancer epithelial/stromal (E/S) ratio, PSMA, CC3 and Ki67 expression. Concordance will be assessed using the Kappa statistic.
Establish a correlation between MRI imaging response and pathologic response | Baseline and mid-treatment (approximately 3 months into treatment)
  MR images will be assessed for response using change in apparent diffusion coefficient (ADC) in order to establish a correlation between imaging response and pathologic response to ADT and EBRT on a lesion-by-lesion basis. Pathologic response will be evaluated as described in Outcome 3. Concordance will be assessed using the Kappa statistic.
Imaging and genomic markers for prostate specific antigen (PSA) recurrence. | Baseline, 3 months post therapy, every 6 months for 5 years
  Determine if imaging and genomic markers that predict for mid-treatment pathologic response also predict PSA recurrence.
Evaluate blood-based biomarkers for treatment response. | Baseline and mid-treatment (approximately 3 months into treatment)
  Messenger RNA from circulating tumor cells (CTCs) will be extracted to determine if presence of androgen receptor variants and a neuroendocrine prostate cancer signature (a score based upon the expression of a set of genes) is correlated with pathologic response (determined as outlined in Outcome 3).

OTHER OUTCOMES:
Changes in cancer gene expression during therapy | Baseline and mid-treatment (approximately 3 months into treatment)
  Evaluate changes in gene expression from pre- to mid-treatment, and their association with response to therapy.
Prognostic significance of higher order radioman metrics | Baseline and mid-treatment (approximately 3 months into treatment)
  Higher order radiomic metrics (e.g. measures of PET lesion heterogeneity obtained using open-source radiomic software) will be assessed as potential predictive markers for pathologic treatment response (measured as outlined in Outcome 3) to ADT and EBRT.

CONTACTS AND LOCATIONS:
Overall Officials: John Floberg, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No